CLINICAL TRIAL: NCT04704167
Title: Comparison of 3D Titanium Miniplates Versus 3D Titanium Mesh Tray as a Method of Fixation for Double Barrel Vascularized Fibular Graft for Mandibular Reconstruction: Randomized Clinical Trial.
Brief Title: 3D Titanium Miniplates Versus 3D Titanium Mesh Method of Fixation for Double Barrel Vascularized Fibular Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hussam Ashraf Mahmoud Okba, PhD Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMFS3-3-17
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fixation of Double Barrel Vascularized Fibula
Keywords: mandibular reconstruction; double barrel vascularized fibula; 3d plate; 3d titanium mesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D titanium mesh tray (Active Comparator): 3D titanium mesh tray as a method of fixation for double-barrel vascularized fibula
  Interventions: Other: fixation of double barrel vascularised fibula
- 3D titanium miniplate (Experimental): 3D titanium miniplate as a method of fixation for double-barrel vascularized fibula
  Interventions: Other: fixation of double barrel vascularised fibula

INTERVENTIONS:
Other: fixation of double barrel vascularised fibula — 3D titanium miniplate or 3D titanium mesh tray are used as a method of fixation for double barrel vascularized fibula

SUMMARY:
The double barrel fibula flap presents many advantages such as adequate, constant geometry, proper dimensions for implant placement, double periosteal and medullary blood supply allowing multiple osteotomies, correct contouring, an adequate pedicle length and low donor site morbidity. Bone thickness, height and its bi-cortical structure seem to be ideal for long-term implant prosthetic rehabilitation. Fixation of double barrel fibula could be done using 3D titanium mini-plate which offers a low profile, less hardware and less chance to remove for later implant placement. Aim of the study is to compare the efficiency of fixation double barrel vascularized fibular graft for mandibular reconstruction using 3D miniplate versus 3D titanium mesh tray

DETAILED DESCRIPTION:
Aim of the study is to compare the efficiency of fixation double barrel vascularized fibular graft for mandibular reconstruction using 3D miniplate versus 3D titanium mesh tray

Hypothesis:

Null hypothesis: There is no difference in the clinical and radio graphical parameters between 3D miniplate fixation versus a 3D titanium mesh tray fixation of double barrel vascularized fibular graft.

If the results are significant (i.e. results are unlikely to be explained by chance alone), the null hypothesis is rejected.

Primary objective: to evaluate bone height changes for double barrel vascularized fibular graft after mandibular reconstruction.

Secondary objective: to evaluate volumetric bone changes for double barrel vascularized fibular graft after mandibular reconstruction.

monitoring success of double vascularized fibular graft in mandibular reconstruction.

Trial design:

* Randomized clinical trial
* A trial will be carried out by a research in Oral &Maxillofacial Surgery department and Ahmed Maher Hospital
* Equal randomization: participants with equal probabilities for intervention and allocation and ratio 1:1.
* Positive controlled: Both groups receiving treatment.
* Parallel group study: Each group of patients receives a single treatment simultaneously.

Preoperative phase:

Patients will be subjected to:

* Case history including personal data, medical, surgical and family history.
* Clinical examination.
* Multi-Slice Computed tomography (CT) for mandible.
* Measuring the defect size
* Computed angiography for the lower limbs.
* Preoperative anaesthesia assessment for fitness for general anaesthesia.
* A Foot Allen Test9
* A stereolithographic model for the patient mandible with reconstructed with double barrel vascularized fibular graft will be printed.

Operative Phase:

* Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
* Apron incision in neck is done in usual manner
* Exposure of neck vessel (external carotid artery and external jugalr vein and their branches)
* Harvesting fibula in usual manner.
* Splitting the fibula to increase its vertical height using double barrel technique and follow planned mandibular contour.
* Fixing the harvest fibula flap to the remaining mandible with reconstruction plate.
* Fixing the top part of the harvested fibula with 3D titanium miniplate or 3D titanium mesh tray (0.6 mm thickness).
* Anastomosing the peroneal artery and vein with the corresponding neck artery and vein
* The remaining flexor halluces longus muscle is sutured to the tibialis posterior muscle and to the interosseous membrane to help preserve great toe flexion.
* A suction drain may be placed between the muscles exiting the inferior limit of the skin incision.
* Closure of skin incision of neck and lower limb in usual manner and placement of drains.

Post-operative phase:

Post-operative medication:

* Amoxicillin/Clavulanic acid 1.5 gram vial injection every 12 hour for 5 days
* Diclofenac Potassium 75mg ampoule Intramuscular injection every 12 hour for 5 days
* Corticosteroids injection for the first 2 days.
* Anticoagulant Subcutaneous injection for 5 days

Post-operative wound care:

* Evaluate suction drains daily and remove them only when <30 mL of serum is collected within a 24 h period.
* Adequate compression is provided by circumferentially wrapping the leg with a compressive, but not too tight, dressing.

No ambulation is allowed within the first 2 weeks. Upon ambulation, partial weightbearing is begun with the aid of crutches followed by full weight bearing ambulation

. Recruitment:

* Patients will be selected by the supervisors and the researcher from outpatient clinic of Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Cairo University- and Ahmed Maher Hospital.
* Screening of patients will continue until the target population is achieved.
* Identifying and recruiting potential subjects is achieved through patient database.

B) Assignment of interventions

Allocation:

Randomization:

The total sample size n= will be calculated and the sample sizes in each group will be pre-specified exactly and are under the direct control of the investigator.

1. Method of random sequence generation: (computerized random number generator).
2. Allocation ratio: (1:1).
3. Type of randomization: simple

Allocation concealment mechanism:

cards will take the generated sequence numbers one number for each card then these cards will be placed within opaque sealed envelopes. Then these Envelops will be placed in a container (box), each participant will grasp one envelop blindly during the preoperative preparation.

Implementation Senior supervisor (EH) is the person who will generate the allocation sequence. Principal investigator (HO) will enroll the participants and assign the participants for intervention.

Masking/blinding:

Because the two interventions used in this trial are easily recognized by the participants and the investigator, neither the investigator (HO) nor the participant can be blinded. But the statistician will be blinded.

C) Data collection, management, and analysis:

Data collection methods (HO) who will be responsible for outcomes assessment. Information on demographic data and past and concurrent medical history was obtained by interviewing the patient.

During Visit 1 (T1 Surgery day), Data regarding personal information, operative procedure (including surgical procedure- intraoperative complications- operation time) and postoperative complication will be recorded each in the specified section in prepared form. At (T2 one week postoperatively) follow-up scheduled for stitch removal and any complications also will be recorded. In the visit 3&4 (T3 & T4 at 3& 6months) patient will be recalled for routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient who require mandibular resection due to tumor, trauma, osteomyelitis or osteoradionecrosis.
* Patient with Mandibular defect >6 centimeter (cm).

Exclusion Criteria:

* • Patients with systemic condition counteracting with the surgical procedure.

  * Patients with conditions contraindicating fibular flap.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
bone height changes for the double barrel vascularized fibular graft | 6 months
  measure bone height changes for the double barrel vascularized fibular graft

SECONDARY OUTCOMES:
volumetric bone changes for the double barrel vascularized fibular graft | 6 months
  measure volumetric bone changes for the double barrel vascularized fibular graft
monitoring viability of the double barrel free vascularized graft | 2 weeks
  monitoring viability of the double barrel free vascularized graft

CONTACTS AND LOCATIONS:
Overall Officials: Hussam A Okba, master, Principal Investigator — Cairo University faculty of dentistry
Locations (1):
- Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD will be shared